CLINICAL TRIAL: NCT03089333
Title: Effects of Dapagliflozin, an SGLT2 Inhibitor, on Hemodynamic Parameters, Target Organ Damage and Obesity Profile in Resistant Hypertensive Subjects
Brief Title: Effects of SGLT2 Inhibitor on Hemodynamic Parameters in Resistant Hypertensive Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Rodrigo Modolo, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016004830
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2; Blood Pressure; Obesity; Cardiac Hypertrophy; Microalbuminuria; Vascular Stiffness
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Obesity; Cardiomegaly | interventions — dapagliflozin; Glyburide; Tablets

STUDY DESIGN:
Intervention Model Description: Two-way crossover design
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10mg daily for 12 weeks.
  Interventions: Drug: Dapagliflozin 10mg; Drug: Glibenclamide 5Mg Tablet
- Glibenclamide (Active Comparator): Glibenclamide 5mg daily for 12 weeks.
  Interventions: Drug: Dapagliflozin 10mg; Drug: Glibenclamide 5Mg Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin at a dose of 10mg daily in combination with metoformin and current antihypertensive therapy for 12 weeks
  Other Names: FARXIGA®
Drug: Glibenclamide 5Mg Tablet — Glibenclamide at a dose of 5mg daily in combination with metoformin and current antihypertensive therapy for 12 weeks
  Other Names: Glibenclamide

SUMMARY:
New strategies trying to achieve blood pressure control and consequently reduce cardiovascular risk in resistant hypertensive subjects are promising. In this context, the SGLT2 inhibitor dapagliflozin, not yet investigated in resistant hypertension, arises as a potential drug in order to impact on blood pressure levels, as well as target organ damage and adiposity in this high-risk population.

DETAILED DESCRIPTION:
Objective: The investigators aim to assess whether the intervention with the SGLT2 inhibitor -dapaglifozin - reduces PA levels, target organ damage, fat profile and change the adipokines levels in patients with resistant hypertension with DM2. Methods and design: This crossover randomized, double-blind, interventional study controlled by standard therapy will include 20 patients with resistant hypertension and type 2 diabetes, followed in Outpatient Clinic specialized in Resistant Hypertension at clinical Hospital-UNICAMP. They will be randomly assigned into two groups (1) initially treated with dapagliflozin in combination with their usual antihypertensive therapy and metformin, at 12 weeks (n = 10) or group (2) Control initially treated with glibenclamide at a dose of 5mg daily in combination with antihypertensive therapy usual and metformin, at 12 weeks (n = 10). Office ambulatory and home BP measurements; anthropometric measurements, determination of vascular stiffness by pulse wave velocity, echocardiogram, body bioimpedance, enzyme immunoassays for the determination of adipokines, and lab tests to evaluate biochemical parameters will be performed pre- and after the use of both treatments. Glycemic parameters, and weight will be assessed every 4 weeks. Results and conclusion: The use of SGLT2 inhibitor in these patients may provide new strategies for treatment of patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertension and type 2 diabetes diagnoses after a 6-month follow-up
* Use of metformin therapy
* Therapy adherence
* Agree to participate in the research protocol and sign the informed consent form

Exclusion Criteria:

* secondary Hypertension
* pseudoresistance hypertension (poor medication adherence and white coat hypertension)
* patients with symptomatic ischemic heart disease, impaired renal function, liver disease and history of stroke, myocardial infarction and peripheral vascular diseases
* pregnancy
* smoking
* autoimmune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline and 12 weeks
  Change in Office Systolic Blood Pressure after 12 weeks of treatment

SECONDARY OUTCOMES:
Change in Ambulatory Systolic Blood Pressure | Baseline and 12 weeks
  Change in Ambulatory Systolic Blood Pressure after 12 weeks of treatment
Change in weight | Baseline and 12 weeks
  Change in body weight
Change in arterial stiffness | Baseline and 12 weeks
  Change in arterial stiffness measured by Sphygmocor device
Change in left ventricular hypertrophy | Baseline and 12 weeks
  Change in left ventricular hypertrophy measured by Echocardiogram
Change in microalbuminuria | Baseline and 12 weeks
  Change in microalbuminuria measured by Urine Albumin/Creatinine Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Modolo, MD, PhD, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas (UNICAMP), Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided